CLINICAL TRIAL: NCT03768674
Title: English Title: Extreme Challenges - Psychopathology, Treatment Organization and Experiences Among Psychiatric Inpatients With Severe Self-harming Behavior in Norway
Brief Title: Extreme Challenges - Psychopathology & Treatment Experiences Among Severly Selfharming Inpatients in Norway
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Extrastiftelsen (Other); National Advisory Unit for Personality Psychiatry (NAPP) (Unknown); Research Group Personality Psychiatry (Unknown); Network for personality-focused treatment (Unknown); National Centre for Suicide Research and Prevention (NSSF) (Unknown); Regional Centre for Violence and Traumatic Stress (RVTS) (Unknown); Regional Centre for Early Intervention Psychosis (TIPS SØrØst) (Unknown); Regional collaborators and users (Unknown)
Responsible Party: Principal Investigator, Elfrida H Kvarstein, Head senior consultant/Associate Professor, Oslo University Hospital
Other Study IDs: 2019/FO244009; 2018/1124 (Other: Regional Ethics Committee)
Record Dates: First submitted 2018-11-11; First posted 2018-12-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Self Harm; Personality Disorders; Psychosis; Developmental Disorder; PTSD; Cognitive Impairment
Keywords: Selfharming behaviors
MeSH Terms: conditions — Self-Injurious Behavior; Personality Disorders; Psychotic Disorders; Developmental Disabilities; Stress Disorders, Post-Traumatic; Cognitive Dysfunction | interventions — Functional Status; Health Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatient cohort (Target group): Inpatient at mental health centre/ psychiatric hospital due to severe self-harm. Duration > 4 weeks and/or > five admissions last year.
  Assessment of diagnoses, functioning and health services
  Interventions: Other: Assessment of diagnoses, functioning and health services
- Outpatient comparison cohort: Admitted to treatment within Norwegian Network of personality-focused treatment during 2017-2018.
  Assessment of diagnoses, functioning and health services
  Interventions: Other: Assessment of diagnoses, functioning and health services

INTERVENTIONS:
Other: Assessment of diagnoses, functioning and health services — Systematic differential diagnostics, assessment of psychosocial and personality functioning and treatment/ health services

SUMMARY:
Patients who self-harm are a heterogeneous population. Outpatient treatments structured for borderline personality disorder are often recommended and hospitalization kept to a minimum. However, few studies have focused on the most severe, complex conditions with extreme suicide risk. A recent national investigation from Norway (2017) demonstrated a far larger cohort of extensively hospitalized inpatients with extreme self-harming behaviors than was expected (N=427) - identified in all health regions. Reported challenges were high-risk situations, severe medical sequelae, difficult collaborations across services, and uncertainty about psychiatric diagnoses.

Severe, often bizarre, self-harm is thus a major challenge for both patients and health services. In hospitals, safety measures can involve restrictions and involuntary regimes. As research on this target population is sparse, the current project seeks further understanding of complex conditions - psychopathology, treatment experiences and service collaboration.

The project is a national, multi-center cooperation including patients in psychiatric hospitals in all health regions. It is cross sectional. Data is based on diagnostic interviews, patients' self-reported symptoms and both patients and service providers treatment experiences. The inclusion period for inpatients (N=300) and a comparison sample of outpatients (N=300) is one year.

The target group is inpatients with extreme hospitalization and severe self-mutilation. A comparison group is patients with personality pathology attending outpatient treatments. Recruitment is across health regions.

Aim 1: Investigate psychopathology of patients in the target population and compare to a clinical sample admitted to outpatient treatment

Aim 2: Investigate personality functioning in the target population and compare to a clinical sample admitted to outpatient treatment

Aim 3: a) Investigate health service use in the target population and compare to a clinical sample admitted to outpatient treatment.

b) Investigate treatment experiences and health service collaborations in the target population.

The project will provide rational for future preventive treatment interventions

DETAILED DESCRIPTION:
Design: A cross-sectional investigation. The inclusion period will be one year.

The target group: Patients admitted to inpatient units (adult psychiatry, mental health centres or hospitals) due to risk of severe self-harm. The duration of admissions are either more than 4 weeks and/or patients have had more than five admissions in the preceding year.

The comparison group is a collaboration with the Norwegian Network of personality-focused treatments and includes clinical data from 19 outpatient units within specialist mental health services across Norway (baseline data for 300 patients admitted to treatment during 2017-2018).

Sample size: An inclusion of N=300 patients in the target Group and comparison group

Assessments: The assessment battery combines therapist administered interviews and patient self-report measures to provide a broad differential-diagnostic evaluation and information about treatment and health-service collaborations. It also includes therapist-reports.

Psychopathology: Assessment of psychiatric disorders includes interviews for symptom disorders (MINI), personality traits and disorders (SCID-5-PD, and observer-evaluated global functioning (GAF) administered in both the target and the comparison group. Assessment of the target group will additionally include a screening interview on cognitive functioning (Hayes Ability Screening Index, HASI, specific approval has been given), self-report screening of autism (Ritvo Autisme Asperger Diagnoseskjema - Revidert RAADS-R), and a detailed interview on psychosis (questions from MINI plus).

General, social and personality functioning: The assessment battery includes a combination of well-established, (no cost) self-report measures covering overall functioning, symptoms, trauma, personality functioning and maladaptive behaviors. These will be administered in both the target and the comparison group. More details on assessment battery can be given on request to PI.

Self-harming behaviors: Self-report on self-harming behaviors and suicide attempts last 6 months are included. Assessment of the target group will additionally include a more detailed interview of self-harming behaviors adapted for Norwegian studies (Lifetime Para suicide Count).

Service use, treatment experiences, and health service collaborations: Assessment of previous treatments, age first time, and contact with child/adolescent psychiatry (self-report, both the target and the comparison group), and a detailed interview on medication, treatments, primary health care and welfare services last 6 months (specially designed interview, both target and comparison group). In addition, for the target group, questions about involuntary and restrictive regimes, treatment involvement, confidence, alliance and collaboration within and across health services are included (patient and therapist reported).

Research collaborators:

The PhD candidate will follow the PhD educationary program at the University of Oslo. Main supervisor is also Principle Investigator (E.H.Kvarstein), and co supervisor (G.Pedersen) heads the Network collaboration. The PhD candidate will join the national project group and be an associated member of the Research group for Personality Psychiatry.

The national project group is central in all phases; design, preparations, implementation procedures, evaluation, and presentations of results. It covers all health regions, relevant research environments, clinicians and users. It includes: Middle HR: T.Torgersen, PhD, Western HR: T.Tveit, MD. Southeastern HR: P.A.Ringen, PhD, P.Danielsen, MA, C.A.Sveen (MA), Tore Buer (MD). Northern HR: H.Tvete, MD, T.Høifødt, PhD. National Centre, Suicide Research and Prevention: F.Walby,MA, R.K.Ramleth, MD (BUP). Regional Centre, Violence and Traumatic Stress: I.Lunde, MA. Early intervention Psychosis: K.L.Romm, PhD. Personality Psychiatry National Advisory Unit: Ø.Urnes,MD. User experience: T.Røstbakken, M.Pettersen, A.Holst.

The Research group for personality psychiatry (University of Oslo/Oslo University Hospital) is an active, well-established research group with engagement in national and international research collaborations specializing on personality pathology and clinical research.

The principle investigator (PI) and main supervisor of this project, E.H.Kvarstein, associate professor, University of Oslo/ Head senior consultant, Section for Personality Psychiatry, Oslo University Hospital, is head of the Research group of personality psychiatry.

The Norwegian Network for personality-focused treatment is a well-established collaboration aiming to ensure clinical quality, systematic treatment evaluation and generate data for clinical research (anonymous data collection). The Network was established in 1993 and currently includes 19 outpatient treatment teams across Norway for patients with personality disorder. Approximately 400 patients are admitted to treatments within the Network each year (mean treatment duration: 2 years). The Network provides systems for patient assessment and progress evaluation, systematic feedback reports on clinical outcomes and supervision/seminars on diagnostic assessment and treatment. The main (ongoing) research project in the Network is a multi-centre feasibility investigation of evidence-based treatment for personality disorder (started in 2017) aiming to include longitudinal treatment data for 500 patients.

"Extreme challenges" is a research collaboration between the national project group and the Network. Baseline data from the multi-centre project constitute the outpatient comparison group in "Extreme challenges" (300 patients, admitted to outpatient treatment in 2017-18, data available in 2020).

Cosupervisor in the PhD project, head of the Network, is senior researcher Geir Pedersen. He is affiliated within the Section for Personality Psychiatry, Oslo University Hospital and the University of Oslo. He is a member of the research group.

Norwegian National Advisory Unit on Personality Psychiatry (NAPP) is the initiator of the current project and the organizer of the national project group. With the establishment of an expert user panel (recruiting users from the whole country), NAPP has also had an active role establishing user engagement in this project.

Plan for activities - practical implementation of the cross sectional investigation: The national project group has already completed a preliminary screening investigation, first publication, and designed the current project. The project group is currently preparing practical implementation of the project (mobilizing regional collaborators, local resource groups and finalizing ethic approvals and systems for data collection).

2018/19: Preparation: Regional preparatory seminars for local clinicians and all collaborators are scheduled to autumn 2019.

2019/2020: Data collection: Assessments of the target population will be performed at the inpatient institutions by local clinicians qualified for diagnostic procedures. During the data collection possibilities for feedbacks/clinical discussion of individual cases will be offered.

Assessments in the comparison group involve measures already implemented (from June 2017).

2021: Dataanalysis, discussion and presentation of results: Datacollection will be concluded and analyses of results proceeds.

2022: Project conclusion

Plan for dissemination of results:

Running information about the project with Norwegian summaries, key researchers and references to all publications will be available at the internet home site of the Research group for Personality Psychiatry in all phases of the project.

Three research publications are scheduled. Manuscripts will be submitted to international peer reviewed journals (open access publication). Research results will also be presented in relevant international/national conferences

When the project is concluded, the project group will arrange a conference for participating clinicians/institutions/organizations, evaluating the investigation, implications and further developments.

User involvement:

The project-group includes three members with relevant user experience, Thea Røstbakken, Mona Pettersen and Andrea Holst.

Ethical considerations The regional ethical committee (REC) has approved the investigator's application for ethical approval. REC reference number is: 2018/1124 A (REC South East).

ELIGIBILITY:
Inclusion Criteria Target population:

* Admitted to inpatient units (adult psychiatry, mental health centres or hospitals) due to risk of severe self-harm.
* Duration of admissions either > 4 weeks and/or > five admissions preceding year.

Exclusion Criteria Target population:

• Not inpatients at a psychiatric, adult (18-60 yrs) institution

Inclusion Criteria comparison population:

• Assessed for outpatient treatment within the outpatient Network

Exclusion criteria comparison population:

• Assessed but not admitted to outpatient treatment within the Network

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The target population is patients with extensive hospitalization due to selfharming behaviors
Sampling Method: Probability Sample
Enrollment: 1640 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Psychiatric Disorders as assessed by M.I.N.I.plus | 2019-2021
  Diagnoses will be assessed by use of semistructured clinical interview: Mini International Neuropsychiatric Interview (M.I.N.I plus)
Post Traumatic Stress Disorder as assessed by PTSD CL 5 | 2019-2021
  Presence and severity of PTSD symptoms will be assessed by PTSD Checklist for DSM-5 (PTSD CL 5)
Severity of psychiatric symptoms as assessed by PHQ | 2019-2021
  Severity of symptoms will be assessed by patient-reports based on the Patient Health Questionairre (PHQ)
Screening for substance use disorder as assessed by AUDIT/DUDIT | 2019-2021
  Additional screening for substance abuse by self-report Alcohol/Drug use disorder identification test (AUDIT/DUDIT)
Personality Disorders as assessed by SCID 5 PD | 2019-2021
  Diagnoses will be assessed by use of the Structured Clinical interview for Diagnoses of Personality Disorders according to DSM-5: SCID-5-PD
Psychosocial functioning I as assessed by GAF | 2019-2021
  Global functioning will be assessed by use of the observer-rated Global assessment of functioning (GAF)
Psychosocial functioning II as assessed by WSAS | 2019-2021
  Global functioning will be assessed by use of self-report: WOrk and Social adjustment Scale (WSAS)
Learning disability screening as assessed by HASI | 2019-2021
  Learning disability will be assessed by use of Hayes Ability Screening Index (HASI)
Autism spectrum screening as assessed by RAADS-R | 2019-2021
  Screening for autism will entail use of The Ritvo Autism Asperger Diagnostic Scale-Revised (RAADS-R)
Overall personality functioning as assessed by SIPP-118 | 2019-2021
  Assessment of personality functioning entails use of the Severity Indices for Personality Functioning (SIPP-118)
Emotional regulation as assessed by DERS | 2019-2021
  Assessment of problems with emotional dysregulation entails use of Difficulties in emotional regulation scale (DERS)
Aggressive behaviors as assessed by MOAS | 2019-2021
  Assessment of problems with aggressive outbursts or behaviors will be assessed by Items from the Modified Overt Aggression Scale (MOAS)
Alexithymia as assessed by TAS-20 | 2019-2021
  Assessment of aspects of affect consciousness will be assessed by the Toronto Alexithymia scale (TAS-20)
Close relationships and attachment patterns as assessed by ECR | 2019-2021
  Assessment of capacities and maladaptive patterns in close relationships will be assessed by the inventory: Experiences in close relationships (ECR).
Selfharming behaviors as assessed by LPC | 2019-2021
  Detailed assessment of selfharming behaviors will entail use of the interview: Lifetime Para suicide Count (LPC)
Specialist mental health service utilization I as assessed by specific interview | 2019-2021
  Interview designed for this project for systematic assessment of the volume of service use last six months (number of outpatient consultations).
Specialist mental health service utilization II as assessed by specific interview | 2019-2021
  Interview designed for this project for systematic assessment of the volume of service use last six months (number of inpatient (hospital) admissions).
Specialist mental health service utilization III as assessed by specific interview | 2019-2021
  Interview designed for this project for systematic assessment of the volume of service use last six months (number of inpatient days in hospital).
Specialist mental health service treatment as assessed by specific interview | 2019-2021
  Interview designed for this project for systematic assessment of type of treatment (category) received last six months.
Welfare services as assessed by specific interview | 2019-2021
  Interview designed for this project for systematic assessment of type of welfare service (category) last six months.
Age at first contact with specialist mental health services as assessed by specific interview | 2019-2021
  Age (years) at first contact with mental health services

CONTACTS AND LOCATIONS:
Overall Officials: Elfrida H Kvarstein, MD,PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03768674/Prot_000.pdf